CLINICAL TRIAL: NCT04642833
Title: Incidence and Clinical-pathological Characteristics of Prostate Cancer in Kidney Transplants Recipients ( KTRs)
Brief Title: Prostate Cancer in Renal Transplants Recipients
Acronym: RENPRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Florence (Other)
Collaborators: Giandomenico Roviello (Unknown); Pietro Spatafora (Unknown); Graziano Vignolini (Unknown); Sergio Serni (Unknown); Simone Caroassai (Unknown); Gabriella Nesi (Unknown)
Responsible Party: Principal Investigator, Donata Villari, Researcher, University of Florence
Other Study IDs: DVillari
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer; Renal Transplantation; Kidney Transplant Recipients
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Kidney transplantation is considered the standard of care for patients with end-stage kidney disease under chronic dialysis treatment. Today, modern surgical techniques have dramatically improved the quality of life and the overall survival of renal transplant recipients (RTRs) . Besides, the use of novel immunosuppressors have increased the 1-year graft survival rate and decreased acute rejection rate . Unfortunately, several transplantation-related diseases including cancer, cardiovascular disease and infection may affect the survival of renal transplant recipients. It has been estimated that RTRs are 2- to 5- fold more likely to develop cancer compared to the general population. Therefore, the development of cancer has become a major concern as it is currently one of the main causes of death in RTRs. The increasing incidence of post-transplant malignancies is generally attributed to immunosuppression which leads to impaired immunosurveillance of cancer cells and virals infections capable of cancer development. Additionally, it has been observed a direct and specific pro-oncogenic effect on RTRs of immunosuppressive drugs and other immunosuppression-independent factors such as the increased age of RTRs, the male gender and the pre-transplant dialysis duration . Prostate cancer is the second most diagnosed cancer in men and the most common non-skin solid neoplasm in RTRs. Generally, the vast majority of post kidney transplantation prostate cancers are localised; however, due to the lack of randomized studies, no specific guidelines for the management of localized prostate cancer are available and, consequently, RTR patients are being treated with surgery or radiotherapy according to national or local guidelines. The concomitant use of immunosuppressors and the presence of the kidney graft in the pelvic cavity make the treatment of localised prostate cancer post kidney transplantation more challenging, highlighting the need for these patients to be addressed to urological oncology centres with surgeons familiar with oncological and transplant surgery.

Prostate cancer is the second most diagnosed cancer in men and the most common non-skin solid neoplasm in RTRs, however, little studies describe the real incidence of prostate cancer in RTRs.

The aim of this study is to retrospectively review a 25-year experience at the Florence Transplant Center in order to evaluate the incidence of prostate cancer and its possible clinical/pathological factors able to influence the survival.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing kidney transplantation in the period from July 1991 to September 2016
* Development of prostate cancer confirmed histologically
* Written informed consent

Exclusion Criteria:

• Lack of clinical and prognostic data on selected patients

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by prostate cancer after kidney transplantation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-01-18 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
To investigate the incidence of prostate cancer in patients who underwent to renal transplantation from July 1991 to September 2016 | 15 months

SECONDARY OUTCOMES:
To retrospectively evaluate possible clinical/pathological factors able to influence the survival of prostate cancer in RTRs | 15 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florence, Florence, Italy